CLINICAL TRIAL: NCT04370613
Title: Imagery Vividness and Arousal Responses to Prospective Imagery
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-06507
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Mental Imagery; Skin conductance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Prospective Imagery visualization task — Participant visualizes brief mental imagery of prospective situations of different valence (neutral, positive, negative).

SUMMARY:
Research has shown that mental imagery appears to carry emotion better than verbal communication. One way this can be noted is that emotional mental imagery trigger physiological arousal responses. These may be important for treatment techniques using mental imagery, such as imaginal exposure and imagery re-scripting. However, as the development of clinical applications increasingly considers the use of flashpoint imagery, i.e. mental imagery of short duration, it is of interest to examine whether also flashpoint imagery trigger arousal responses. This study examines the arousal response to flashpoint imagery of different valence (positive, negative, and neutral).

Moreover, emerging evidence suggest that depressed individuals find it more difficult to produce mental imagery of positive future events (less accessible and vivid) than healthy controls. In addition, individuals with clinical anxiety appear to be able to produce imagery of negative future events more easily than healthy controls. This study explores whether these results can be noted also in sub-clinical symptoms of depression and anxiety, and if so, if they are accompanied with corresponding changes in arousal responses.

DETAILED DESCRIPTION:
This study takes part in a single session. Participants will produce flashpoint imagery of future events while skin conductance responses, imagery vividness ratings, valence and arousal ratings are collected. Participants will also fill in questionnaires on depression and anxiety symptoms, as well as a questionnaire measuring general propensity for mental imagery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Fluent in Swedish
* Willing and able to provide informed consent and complete study procedures

Exclusion Criteria:

* Current psychiatric disorder
* Current use of psychotropic medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Imagery vividness ratings | Day 1
  Scale: 1-5; no image at all - image as clear and vivd as real life
Skin conductance response (SCR) | Day 1
  SCR is used to measure physiological arousal response to the mental imagery production. The study evaluates differences in SCR between valences of prospective imagery (neutral, negative, positive) and possible covariation with self-rated anxiety or depression symptoms.

SECONDARY OUTCOMES:
Time in seconds it takes to construct a situation to visualize | Day 1
  Measured as the time period from the presentation of the instruction until the participant reports a constructed situation.
Subjective Valence Ratings | Day 1
  Subjective Valence Ratings for each produced mental imagery (0-100; negative to positive)
Subjective Arousal Ratings | Day 1
  Subjective Arousal Ratings for each produced mental imagery (0-100; 0=no arousal, 100=maximum arousal)
The Vividness of Visual Imagery Questionnaire | Day 1
  This is a self-rated questionnaire measuring vividness of visual mental imagery. Higher scores indicate higher level of vividness (range 0-80)
State-Trait Anxiety Inventory | Day 1
  This is a self-rated questionnaire measuring trait anxiety. Higher scores indicate higher level of trait anxiety (range 20-80)
Formulär för patienthälsa (PHQ-9) | Day 1
  This is a self-rated questionnaire for measuring depression symptoms. Higher scores indicate more symptoms of depression (range 0-27 + specific question of how disabling the symptoms are)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ågren, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Department of Psychology, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data, study protocol, and ICF will be available at Open Science Framework (OSF) upon publication. Statistical analysis plan will be pre-registered at OSF.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available upon publication